CLINICAL TRIAL: NCT00288730
Title: A Randomized, Double-Blinded, Placebo-Controlled Study of Two Doses of NATRECOR hBNP (Nesiritide) Administered as a Continuous Infusion in Subjects With Decompensated CHF
Brief Title: A Study of Two Doses of Intravenous NATRECOR hBNP (Nesiritide) in Patients With Worsening Congestive Heart Failure Who Have Difficulty Breathing at Rest
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005197
Record Dates: First submitted 2006-02-03; First posted 2006-02-08 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Heart Failure, Congestive; Heart Decompensation
Keywords: Heart Failure; Renal Dysfunction; Cardiomyopathy; Heart Decompensation; Dyspnea Paroxysmal
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Cardiomyopathies; Dyspnea, Paroxysmal | interventions — Natriuretic Peptide, Brain

ARMS (1):
- 001 (Experimental): nesiritide
  Interventions: Drug: nesiritide

INTERVENTIONS:
Drug: nesiritide

SUMMARY:
The purpose of this study is to assess the safety and efficacy of two doses of intravenous NATRECORÂ® hBNP (a recombinant form of the natural human peptide normally secreted by the heart) versus placebo in the treatment of patients with symptomatic, decompressed congestive heart failure (CHF).

DETAILED DESCRIPTION:
Human studies reported by SJ Holmes et al, 1993, AM Richards et al, 1993 and M. Yoshimara et al, 1991 show that administration of externally produced hBNP produces vasodilation; antagonism of the hormone system that helps regulate long term blood pressure and blood volume in the body; and an increase in urine output containing large amounts of salt. These studies suggest hBNP may be a potent agent for the treatment of acute congestive heart failure (CHF) with a unique combination of desirable effects on the flow of blood throughout the body; the hormones secreted by the nervous system; and support of copious salt outputs by the renal system not provided by currently available therapies. Plasma hBNP levels are elevated in CHF and hBNP may be one of the body's natural compensatory mechanisms to augment cardiac functions in a failing heart. NATRECOR® hBNP is Scios' proprietary form of hBNP and it is identical to the amino acid sequence in the naturally occurring hormone. This is a randomized, double-blinded, placebo-controlled, multicenter study to determine the efficacy of two distinct doses of NATRECOR® hBNP in patients with symptomatic, decompensated congestive heart failure to decrease pulmonary capillary wedge pressure, as measured by a blinded comparison to placebo after 6 hours of treatment. Patients are randomized to receive either a placebo or one of two doses (0.015 or 0.03 µg/kg/min) of NATRECOR® hBNP. The study hypothesis is that NATRECOR ® hBNP is well tolerated and an effective agent for the short-term management of hospitalized patients with symptomatic, decompensated CHF. Patients are randomized to receive either a placebo or one of two doses (0.015 or 0.03 µg/kg/min) of NATRECOR® hBNP. Doses are administered one time only, an intravenous loading bolus, followed by continuous intravenous infusion for 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic congestive heart failure (CHF)
* symptomatic, decompensated CHF for which intravenous therapy is deemed appropriate for the hospitalized patient
* documentation of pulmonary capillary wedge pressure (PCWP) >= 18 mm Hg, Cl <= 2.7 mL/min/m² and systolic blood pressure >= 90 mm Hg with consistent baseline hemodynamic measurements.

Exclusion Criteria:

* Had a myocardial infarction within the previous 48 hours or unstable angina
* stroke within the previous 3 months or other evidence of significantly compromised central nervous system perfusion
* has significant valvular stenosis hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, biopsy-proven active myocarditis, or complex congenital heart disease
* receiving ongoing treatment with an intravenous vasostrictive agent for this episode of decompressed CHF that could not be discontinued for an appropriate washout period to permit the reassessment of baseline hemodynamic and clinical status prior to initiating drug study
* clinical status so unstable that the subject can not tolerate placement of a Swan-Ganz catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 1996-10; Study Completion 1997-08 (Actual)

PRIMARY OUTCOMES:
Hemodynamic effects assessed by an increase in cardiac output without an increase in heart rate, measured at 1.5, 3, 4.5 and 6 hours.

SECONDARY OUTCOMES:
Hemodynamic improvements sustained throughout at least 24 hours of infusion: improvements in overall clinical status and specific signs and symptoms of CHF after 6 hours of treatment; reduction in plasma aldosterone levels.

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- [Result] Mills RM, LeJemtel TH, Horton DP, Liang C, Lang R, Silver MA, Lui C, Chatterjee K. Sustained hemodynamic effects of an infusion of nesiritide (human b-type natriuretic peptide) in heart failure: a randomized, double-blind, placebo-controlled clinical trial. Natrecor Study Group. J Am Coll Cardiol. 1999 Jul;34(1):155-62. doi: 10.1016/s0735-1097(99)00184-9. PMID 10400005